CLINICAL TRIAL: NCT02717689
Title: A Randomised Pragmatic Trial Of Corticosteroid Optimisation In Severe Asthma Using A Composite Biomarker Algorithm To Adjust Corticosteroid Dose Versus Standard Care
Brief Title: A Pragmatic Trial of Corticosteroid Optimisation in Severe Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Medical Research Council (Other Government); Hoffmann-La Roche (Industry); Aerocrine AB (Industry)
Responsible Party: Principal Investigator, Liam Heaney, Professor of Respiratory Medicine, Belfast Health and Social Care Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2016-03-16; First posted 2016-03-24 (Estimated); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Severe Persistent Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biomarker arm (Experimental): Biomarker based adjustment of corticosteroid dose.
  Interventions: Other: Biomarker based adjustment of corticosteroid dose
- Standard care (No Intervention): The subject's corticosteroid dose will be adjusted based upon asthma symptom control and lung function

INTERVENTIONS:
Other: Biomarker based adjustment of corticosteroid dose — The subject's corticosteroid dose will be adjusted based upon biomarker results (FeNO, eosinophils and periostin)
  Arms: Biomarker arm

SUMMARY:
This study explores if a composite biomarker strategy predicts exacerbation risk in patients with asthma on high dose inhaled corticosteroid (+/-long-acting beta agonist) treatment and to evaluate the utility of this composite score to facilitate personalised biomarker specific titration of corticosteroid therapy in this population.

DETAILED DESCRIPTION:
Asthma affects an estimated 300 million people worldwide with a population prevalence of ca 15% in the UK. The WHO has estimated UK disability adjusted life-years per 100,000 population for asthma to be greater than diabetes and breast cancer. Much of this excessive disability is in the 10-20% of patients with asthma which is difficult to control despite currently available therapies. This high morbidity and disproportionate use of health care resources reflects the considerable unmet need in this patient group, and their significance for health care providers.

Asthma has been traditionally 'stratified' on the basis of response to 'step-wise' incremental treatment with inhaled corticosteroid (ICS) therapy forming the cornerstone of this approach. However, more recently, asthma has been stratified on the basis of inflammatory phenotype to better understand disease heterogeneity with a view to developing biomarkers of therapeutic response and for the better targeting of both new and existing treatments.

Investigators have recently examined the predictive value of a composite biomarker strategy using FeNO, blood eosinophils and serum periostin together to predict exacerbation risk in the placebo arms of clinical trials. Investigators propose to examine if this composite biomarker strategy predicts exacerbation risk in patients with asthma on high dose ICS (+/-long-acting beta agonist) treatment and to evaluate the utility of this composite score to facilitate personalised biomarker specific titration of corticosteroid therapy in this population. This study will examine subjects with FeNO<45 ppb and the scoring system will potentially allow identification of a 'low-risk' group who can safely reduce corticosteroid dose. This study will address a second important question of estimating the proportion of patients with severe disease who develop typical (T2)-driven eosinophilic inflammation on progressive corticosteroid withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 80 years at screening visit
2. Able and willing to provide written informed consent and to comply with the study protocol
3. Baseline FeNO< 45 ppb at screening
4. Severe asthma confirmed after assessment by an asthma specialist. Diagnosed with asthma at least 12 months prior to screening
5. Current asthma treatment with LABA plus high doses of inhaled corticosteroids (≥1000 µg FP daily or equivalent)
6. Patients on an ICS/LABA single inhaler strategy must be switched to fixed dosing ICS/LABA for 4 weeks prior to screening
7. Documented history of reversibility of ≥12% change in FEV1 within the past 24 months or during screening period, as demonstrated by:

   * Documented airflow obstruction (forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC ) <70%), where FEV1 has varied by ≥12% either spontaneously or in response to oral corticosteroid (OCS) therapy or bronchodilators either between or during clinic visits Or
   * A 20% drop in FEV1 (PC20) to methacholine <8 mg/mL or a 15% fall in FEV1 (PD15) after inhaling a cumulative dose of mannitol of ≤635 mg indicating the presence of airway hyperresponsiveness. If sites customarily use histamine to perform tests of airway responsiveness, this may be used in place of methacholine.

Exclusion Criteria:

1. Acute exacerbation requiring oral corticosteroids in previous 4 weeks before screening.
2. Known severe or clinically significant immunodeficiency, including, but not limited to, human immunodeficiency virus (HIV) infection.
3. Currently receiving or have historically received intravenous immunoglobulin for treatment for immunodeficiency.
4. If recently commenced on a leukotriene receptor antagonist or theophylline, stable on treatment for 4 weeks prior to screening
5. Known current malignancy or current evaluation for a potential malignancy or history of malignancy within 5 years prior to baseline. With the exception of basal-cell and squamous-cell carcinomas of the skin and carcinoma in situ of the cervix uteri that have been excised and cured.
6. Other clinically significant medical disease or uncontrolled concomitant disease despite treatment that is likely, in the opinion of the investigator, to require a change in therapy or impact the ability to participate in the study
7. History of current alcohol, drug, or chemical abuse or past abuse that would impair or risk the subject's full participation in the study, in the opinion of the investigator
8. Current self-reported history of smoking (including electronic inhaled nicotine products) or former smoker with a smoking history of >15 pack-years

   * A current smoker is defined as someone who has smoked one or more cigarettes per day (or marijuana or pipe or cigar) for ≥ 30 days within the 24 months prior to the screening visit (Day -14) and / or cotinine positive at screening
   * Any individual who smokes (cigarettes, marijuana, pipe, or cigar) occasionally, even if for < 30 days within the 24 months prior to the screening visit (Day -14), must agree to abstain from all smoking from the time of consent through completion of study
   * A former smoker is defined as someone who has smoked one or more cigarettes per day (or marijuana or pipe or cigar) for ≥ 30 days in his or her lifetime (as long as the 30-day total did not include the 24 months prior to the screening visit [Day -14]).
   * A pack-year is defined as the average number of packs per day times the number of years of smoking.
9. Current use of an immunomodulatory/immunosuppressive therapy or past use within 3 months or five drug half-lives (whichever is longer) prior to the screening visit
10. Use of a biologic therapy including Omalizumab at any time during the 6 months prior to the screening visit.
11. Bronchial thermoplasty within prior 6 months of the screening visit
12. Initiation of or change in allergen immunotherapy within 3 months prior to the screening visit.
13. Treatment with an investigational agent within 30 days of the screening visit (or five half lives of the investigational agent, whichever is longer).
14. Female patients who are pregnant or lactating.

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with any reduction in corticosteroid dose | 48 weeks
  Proportion of patients with any reduction in oral or inhaled corticosteroid dose at any point over the 48 weeks of the study

SECONDARY OUTCOMES:
Rate of protocol-defined severe exacerbations per patient per year | 48 weeks
Time to first severe exacerbation from randomisation | 48 weeks
Dose of inhaled steroid at end of study | Week 48
Cumulative dose of inhaled corticosteroid during study | 48 weeks
Proportion of patients on oral corticosteroids at the end of the study | Week 48
Proportion of patients who decline to progress to oral corticosteroids despite composite biomarker score of 2 | 48 weeks
Frequency of hospital admission for asthma | 48 weeks
Change in Asthma Control Questionnaire (ACQ-7) | Week 48
Change in FEV1 (volume) | Week 48
Change in exhaled breath nitric oxide level | Week 48
Change in blood eosinophil count | Week 48
Change in serum periostin levels | Week 48
Change in Asthma Quality of Life Questionnaire (AQLQ) | Week 48

OTHER OUTCOMES:
Exploratory biomarker analysis using whole blood gene expression | 48 weeks
  Blood will be taken for whole blood gene expression
Exploratory serum biomarker analysis | 48 weeks
  Blood will be taken for exploratory serum biomarkers
Exploratory plasma biomarker analysis | 48 weeks
  Blood will be taken for exploratory plasma biomarkers
Exploratory urinary biomarker analysis | 48 weeks
  Urine will be taken for exploratory urine biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Liam Heaney, MBBCh MRCP, Principal Investigator — Queen's University, Belfast
Locations (11):
- United Kingdom (11):
  - Belfast Health and Social Care Trust, Belfast, Northern Ireland
  - Heart of England NHS Foundation Trust, Birmingham
  - NHS Greater Glasgow and Clyde, Glasgow
  - University Hospitals of Leicester NHS Trust, Leicester
  - Royal Brompton & Harefield NHS Foundation Hospital, London
  - University College London Hospitals NHS Foundation, London
  - University Hospitals of South Manchester NHS Trust, Manchester
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Foundation Trust, Nottingham
  - Oxford University Hospitals NHS Trust, Oxford
  - University Hospital of Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDowell PJ, Busby J, Hanratty CE, Djukanovic R, Woodcock A, Walker S, Hardman TC, Arron JR, Choy DF, Bradding P, Brightling CE, Chaudhuri R, Cowan D, Mansur AH, Fowler SJ, Diver SE, Howarth P, Lordan J, Menzies-Gow A, Harrison T, Robinson DS, Holweg CTJ, Matthews JG, Pavord ID, Heaney LG. Exacerbation Profile and Risk Factors in a Type-2-Low Enriched Severe Asthma Cohort: A Clinical Trial to Assess Asthma Exacerbation Phenotypes. Am J Respir Crit Care Med. 2022 Sep 1;206(5):545-553. doi: 10.1164/rccm.202201-0129OC. PMID 35549845
- [Derived] Busby J, Matthews JG, Chaudhuri R, Pavord ID, Hardman TC, Arron JR, Bradding P, Brightling CE, Choy DF, Cowan DC, Djukanovic R, Hanratty CE, Harrison TW, Holweg CT, Howarth PH, Fowler SJ, Lordan JL, Mansur AH, Menzies-Gow A, Niven RM, Robinson DS, Walker SM, Woodcock A, Heaney LG; investigators for the MRC Refractory Asthma Stratification Programme. Factors affecting adherence with treatment advice in a clinical trial of patients with severe asthma. Eur Respir J. 2021 Sep 24;59(4):2100768. doi: 10.1183/13993003.00768-2021. Print 2022 Apr. PMID 34561291
- [Derived] Heaney LG, Busby J, Hanratty CE, Djukanovic R, Woodcock A, Walker SM, Hardman TC, Arron JR, Choy DF, Bradding P, Brightling CE, Chaudhuri R, Cowan DC, Mansur AH, Fowler SJ, Niven RM, Howarth PH, Lordan JL, Menzies-Gow A, Harrison TW, Robinson DS, Holweg CTJ, Matthews JG, Pavord ID; investigators for the MRC Refractory Asthma Stratification Programme. Composite type-2 biomarker strategy versus a symptom-risk-based algorithm to adjust corticosteroid dose in patients with severe asthma: a multicentre, single-blind, parallel group, randomised controlled trial. Lancet Respir Med. 2021 Jan;9(1):57-68. doi: 10.1016/S2213-2600(20)30397-0. Epub 2020 Sep 8. PMID 32916135
- [Derived] Hanratty CE, Matthews JG, Arron JR, Choy DF, Pavord ID, Bradding P, Brightling CE, Chaudhuri R, Cowan DC, Djukanovic R, Gallagher N, Fowler SJ, Hardman TC, Harrison T, Holweg CT, Howarth PH, Lordan J, Mansur AH, Menzies-Gow A, Mosesova S, Niven RM, Robinson DS, Shaw DE, Walker S, Woodcock A, Heaney LG; RASP-UK (Refractory Asthma Stratification Programme) Consortium. A randomised pragmatic trial of corticosteroid optimization in severe asthma using a composite biomarker algorithm to adjust corticosteroid dose versus standard care: study protocol for a randomised trial. Trials. 2018 Jan 4;19(1):5. doi: 10.1186/s13063-017-2384-7. PMID 29301585